CLINICAL TRIAL: NCT01885728
Title: A Randomized, Controlled Study Evaluating the Immune-Modulatory Effects of Perioperative Administration of Arginine Rich Nutritional Supplements With Mass Cytometry in Patient Undergoing Surgery
Brief Title: Immune-modulation Effects of an Arginine Rich Nutritional Supplement in Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin Angst (Other)
Responsible Party: Sponsor-Investigator, Martin Angst, Professor of Anesthesia, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27485
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Immunity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arginine rich nutritional supplement (Active Comparator): 237 ml of an arginine rich nutritional supplement 4 times a day for the five days preceding surgery.
  Interventions: Dietary Supplement: An arginine rich nutritional supplement
- No nutritional supplement (No Intervention): No specific nutritional requirements have to be met in this group.

INTERVENTIONS:
Dietary Supplement: An arginine rich nutritional supplement — Impact is a nutritional supplement formulated with 18 grams of protein per serving and 24 essential nutrients including arginine.
  Other Names: 'Impact' made by Nestle Corporation
  Arms: Arginine rich nutritional supplement

SUMMARY:
The primary objective of this study is to characterize the immune-modulatory effects of arginine-rich nutritional supplements in patients undergoing surgery. Numerical and functional changes of all circulating immune cells will be assessed with mass cytometry.

ELIGIBILITY:
Inclusion Criteria:

1. Colon surgery for cancer
2. Patients ≥ 18 and ≤65 years of age
3. Patients willing and able to sign an informed consent form and Health Insurance and Portability Act (HIPAA) authorization and to comply with study procedures

Exclusion Criteria:

1. Patients on immune-suppressant therapy within the last 6 months (e.g. azathioprine or cyclosporine)
2. Patients pretreated (6 months) or currently on chemotherapy for cancer
3. Patients on radiation therapy (within 6 months)
4. Patients on chronic medication with potential immune-modulatory effects (e.g. daily oral morphine-equivalent intake > 30 mg)
5. Patients with metastatic disease
6. Patients with active infectious disease (within 2 months)
7. Patients with significant metabolic disease (e.g. diabetes type I)
8. Patients with clinically significant organ dysfunction including renal and hepatic dysfunction
9. Patients with significant cardiovascular and respiratory comorbidities resulting in impaired function and frailty
10. Patients with autoimmune disease (e.g. lupus)
11. Patients with Hx of substance abuse (e.g., alcoholism, drug dependency)
12. Undernourished patients as indicated by a weight loss >10% during the last 6 months
13. Patients with galactosemia
14. Patients who had undergone previous major abdominal surgery
15. Participation in another clinical trial of an investigational drug or device within the last 30 days prior to the first day of study that, in the investigator's opinion, would create increased risk to the participant or compromise the integrity or either study
16. Pregnancy
17. Other conditions compromising a participant's safety or the integrity of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes in fractional representation of myeloid-derived suppressor cells (MDSC) from baseline. | Base line (prior to 1st administration of arginine supplement), immediately prior to surgery, 24 hours, 72 hours and 120 hours after surgery.
  The fraction of MDSCs will be quantified.
Functional status change of myeloid-derived suppressor cells (MDSC) from baseline. | Base line (prior to 1st administration of arginine supplement), immediately prior to surgery, 24 hours, 72 hours and 120 hours after surgery.
  Intracellular phosphorylation events in MDSCs will be quantified.

SECONDARY OUTCOMES:
Impact of surgery on clinical recovery using multiple clinical measures and a validated questionnaire. | Daily for duration of hospital stay, then every 3 days trough postoperative week 5.
  Outcome measures include the 1) Surgical Recovery Scale, 2) Pain (11-point numerical pain rating scale), 3) Consumption of analgesic drugs.

OTHER OUTCOMES:
Fractional and absolute expansion/contraction of cluster of differentiation 4 (CD4)+ and cluster of differentiation 8 (CD8)+ cells | Base line (prior to 1st administration of arginine supplement), immediately prior to surgery, 24 hours, 72 hours and 120 hours after surgery.
Functional status of cluster of differentiation 4 (CD4)+ and cluster of differentiation 8 (CD8)+ cells | Base line (prior to 1st administration of arginine supplement), immediately prior to surgery, 24 hours, 72 hours and 120 hours after surgery.
Functional potency of cluster of differentiation 4 (CD4)+ and cluster of differentiation 8 (CD8)+ cells | Base line (prior to 1st administration of arginine supplement), immediately prior to surgery, 24 hours, 72 hours and 120 hours after surgery.
Capacity of cluster of differentiation 4 (CD4)+ and cluster of differentiation 8 (CD8)+ cells | Base line (prior to 1st administration of arginine supplement), immediately prior to surgery, 24 hours, 72 hours and 120 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Angst, MD, Principal Investigator — Stanford University SOM
Locations (1):
- Stanford University Hospital, Stanford, California, United States